CLINICAL TRIAL: NCT04974177
Title: A Prospective Observational Study to Determine the Role of Physician Gestalt in Clinical Prediction of COVID-19
Brief Title: A Study to Determine the Role of Physician Gestalt in Predicting COVID-19 in Patients
Status: Completed | Type: Observational
Sponsor: Jubilee Mission Medical College and Research Institute (Other)
Responsible Party: Principal Investigator, SARASWATHY M, Junior Resident, Jubilee Mission Medical College and Research Institute
Other Study IDs: 13/21/IEC/JMMC&RI
Record Dates: First submitted 2021-07-21; First posted 2021-07-23 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: All Patients Undergoing COVID 19 Specific Testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
THIS IS A PROSPECTIVE OBSERVATIONAL STUDY TO DETERMINE THE ROLE OF PHYSICIAN GESTALT IN CLINICAL PREDICTION OF COVID 19.

DETAILED DESCRIPTION:
Among patients attending the Emergency Department, prompt identification of possible cases of COVID 19 is important to avoid the spread. An immediate clinical diagnosis is important for point of care decision making on choice of treatment facility as well as for triaging, testing and to quarantine patients admitted to the hospital from emergency room. Hence this study attempts to find out the role of physician gestalt in early diagnosis and differentiation of COVID 19.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to ED, who undergo COVID 19 specific testing.

Exclusion Criteria:

* Patients with active COVID 19 disease diagnosed outside All brought dead cases. All patients not consenting to take part in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients presenting to ED, who undergo COVID 19 specific testing.
Sampling Method: Non-Probability Sample
Enrollment: 876 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity, positive and negative likelihood ratio of physician gestalt in diagnosis of COVID 19 in patients presenting to ED who are being sent for COVID 19 specific testing. | march 2021- september 2022

SECONDARY OUTCOMES:
Sensitivity, specificity, positive and negative likelihood ratio of clinical and epidemiological variables in patients presenting to ED who are being sent for COVID 19 specific testing. | march 2021- september 2022

CONTACTS AND LOCATIONS:
Locations (1):
- Jubilee Mission Medical College, Thrissur, Kerala, India